CLINICAL TRIAL: NCT02652208
Title: Randomized Trial Comparing Effectiveness of Two Patient Decision Aids for Stable Chest Discomfort
Brief Title: Comparative Effectiveness of Decision Aids for Stable Chest Discomfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Karen Sepucha, Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2014P002292
Record Dates: First submitted 2016-01-08; First posted 2016-01-11 (Estimated); Results first posted 2017-08-29 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Coronary Artery Disease; Stable Angina
Keywords: decision making; decision aids; shared decision making; stable angina; cardiology
MeSH Terms: conditions — Coronary Artery Disease; Angina, Stable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Online decision aid (Active Comparator): This group will receive the access to an online decision aid that covers the main treatment options for stable chest discomfort.
  Interventions: Behavioral: Online decision aid
- Video decision aid (Active Comparator): This group will receive the DVD and booklet decision aid describing stable chest discomfort and the main treatment options including medical therapy and stents.
  Interventions: Behavioral: Video decision aid

INTERVENTIONS:
Behavioral: Online decision aid — The Healthwise online shared decision point for Stable Chest Discomfort
  Arms: Online decision aid
Behavioral: Video decision aid — The Health Dialog DVD and booklet decision aid for Stable Chest Discomfort
  Arms: Video decision aid

SUMMARY:
The purpose of the study is to compare two different types of decision support materials for patients considering treatment for chest pain or chest discomfort from heart disease.

DETAILED DESCRIPTION:
The purpose of the project is to compare the effectiveness of a detailed, video patient decision aid and an online, interactive patient decision aid for treatment of Stable Chest Discomfort. The study will randomly assign eligible participants to receive either the online decision aid or the video decision aid. Participants will complete a survey after reviewing the decision aid that will examine decision quality, use of the intervention, and satisfaction with the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 and older
* English speaking
* Current diagnosis of stable angina
* Ability to access online material and willing to provide an email address

Exclusion Criteria:

* Coronary bypass surgery and/or percutaneous coronary intervention within 6 months
* Diagnosis of unstable angina, acute coronary syndrome, STEMI, non STEMI within 6 months
* Scheduled for nonelective catheterization
* Significant cognitive deficit such that participant is unable to consent for self
* Serious comorbidities or other conditions that make revascularization inappropriate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen R Sepucha, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boden WE, O'Rourke RA, Teo KK, Hartigan PM, Maron DJ, Kostuk WJ, Knudtson M, Dada M, Casperson P, Harris CL, Chaitman BR, Shaw L, Gosselin G, Nawaz S, Title LM, Gau G, Blaustein AS, Booth DC, Bates ER, Spertus JA, Berman DS, Mancini GB, Weintraub WS; COURAGE Trial Research Group. Optimal medical therapy with or without PCI for stable coronary disease. N Engl J Med. 2007 Apr 12;356(15):1503-16. doi: 10.1056/NEJMoa070829. Epub 2007 Mar 26. PMID 17387127
- [Background] Rothberg MB, Sivalingam SK, Ashraf J, Visintainer P, Joelson J, Kleppel R, Vallurupalli N, Schweiger MJ. Patients' and cardiologists' perceptions of the benefits of percutaneous coronary intervention for stable coronary disease. Ann Intern Med. 2010 Sep 7;153(5):307-13. doi: 10.7326/0003-4819-153-5-201009070-00005. PMID 20820040
- [Background] Holmboe ES, Fiellin DA, Cusanelli E, Remetz M, Krumholz HM. Perceptions of benefit and risk of patients undergoing first-time elective percutaneous coronary revascularization. J Gen Intern Med. 2000 Sep;15(9):632-7. doi: 10.1046/j.1525-1497.2000.90823.x. PMID 11029677

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Online Decision Aid | Video Decision Aid
Started | 17 | 17
Completed | 13 | 15
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Online Decision Aid | Video Decision Aid | Total
Number analyzed (Participants) | 13 | 15 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 9
  >=65 years | 7 | 12 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (10.2) | 73 (11.6) | 70 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 9 | 12
  Male | 10 | 6 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 15 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 15 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: Total Knowledge Score
Description: Six multiple choice knowledge items covered important facts patients should know about chest pain or discomfort and treatments. A total knowledge score (0-6) was created by summing the total number of correct responses. A missing knowledge response was marked as incorrect. Any survey with more than three missing knowledge responses did not get a total knowledge score. A higher score indicates higher knowledge on the topic. Both decision aids provided information for answering all knowledge items. Higher knowledge scores are better.
Time Frame: Within 1 week after reviewing the decision aid
Population: All participants who completed and returned a survey within the 6 month study period.
Measure: Mean (Standard Deviation); unit: knowledge score
Arm/Group | Online Decision Aid | Video Decision Aid
Number analyzed (Participants) | 12 | 15
knowledge score | 2.83 (0.72) | 4.0 (1.46)

2. Secondary Outcome: Treatment Leaning (Percentage of Patients Who Have a Clear Treatment Preference)
Description: To determine the percentage of patients who have a clear treatment preference for their stable chest discomfort.
Time Frame: Within 1 week after reviewing the decision aid
Population: Only participants who indicated they currently had symptoms were asked to complete the item
Measure: Count of Participants; unit: Participants
Arm/Group | Online Decision Aid | Video Decision Aid
Number analyzed (Participants) | 6 | 8
Participants | 4 | 5

3. Secondary Outcome: Satisfaction With the Intervention
Description: Number of respondents who rated the material as "very good" or "excellent".
Time Frame: Within 1 week after reviewing the decision aid
Population: All participants who completed and returned a survey within the 6 month study period.
Measure: Count of Participants; unit: Participants
Arm/Group | Online Decision Aid | Video Decision Aid
Number analyzed (Participants) | 13 | 15
Participants | 6 | 10

ADVERSE EVENTS:
Time Frame: Serious and other (not including serious) adverse events were not collected/assessed as part of this survey study
Description: The survey study examining patient reactions to educational materials did not collect adverse event information.
Arm/Group | Online Decision Aid | Video Decision Aid
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes